CLINICAL TRIAL: NCT00036244
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Assess the Efficacy, Safety and Tolerability of RG1068 (Synthetic Human Secretin) in Children With Autism
Brief Title: Synthetic Human Secretin in Children With Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repligen Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RG1068-04
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2005-08-05 (Estimated); Status verified 2005-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Secretin

INTERVENTIONS:
Drug: RG1068 (Synthetic Human Secretin)

SUMMARY:
The purpose of the study is to determine whether multiple doses of secretin are safe and effective in the treatment of children with autism.

ELIGIBILITY:
Autism

Ages: 32 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2002-04; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Southwest Autism Research Center, Phoenix, Arizona
  - UCLA Pediatric Neurology, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - 1st Allergy & Clinical Research Center, Centennial, Colorado
  - Alachua Family Psychiatry, Gainesville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Riley Children's Hospital, Indianapolis, Indiana
  - The Clinical Trials Center:A Division of Children's Hospital, Metairie, Louisiana
  - Hardy Healthcare Associates, Hingham, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - The Ohio State University, Columbus, Ohio
  - Children's Biomedical Center of Utah, Sandy City, Utah
  - Puget Sound Neurology, Edmonds, Washington

REFERENCES:
- See also: Related Info — http://www.repligen.com